CLINICAL TRIAL: NCT00516061
Title: Relationship of Peritoneal Solute Transport Rate With VEGF in Children Undergoing Peritoneal Dialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Other Study IDs: 2006-12-008
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2006-12

CONDITIONS: Peritoneal Dialysis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Vascular endothelial growth factor(VEGF) appears to play a central role in the process leading to peritoneal angiogenesis and increased level of VEGF may contribute to high peritoneal small-solute transport rate (PSTR) in continuous ambulatory peritoneal dialysis (CAPD) patients in adult. In children, lymphatic absorption of solute is greater than adult. VEGF-C is related to lymphogenesis, but its role in peritoneal solute transport rate is not known. In this study, we evaluated possible relationship between dialysate VEGF and VEGF-C levels and PSTR in children.

DETAILED DESCRIPTION:
There was significant correlation between dialysate VEGF165 and VEGF-C levels and significant correlation was noted between dialysate VEGF165 and PSTR. Interestingly, dialysate VEGF-C levels had significant correlation with PSTR. High PSTR seems to be related to elevated VEGF-C and VEGF.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal failure
* children
* peritoneal dialysis

Exclusion Criteria:

* acute illness

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-12; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hoon Paik, M.D., Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea